CLINICAL TRIAL: NCT07303725
Title: Intra-procedural Spectral CT for Image-guided Embolization and Ablation in Interventional Oncology
Status: Recruiting | Type: Observational
Sponsor: Palo Alto Veterans Institute for Research (Other)
Collaborators: Canon Medical Systems, USA (Industry)
Responsible Party: Sponsor
Other Study IDs: KIS0004ARG
Record Dates: First submitted 2025-03-17; First posted 2025-12-26 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-03

CONDITIONS: Liver Cancer (Primary and Metastatic); Renal Cancer
Keywords: spectral CT
MeSH Terms: conditions — Liver Neoplasms; Neoplasm Metastasis; Kidney Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- angiography mapping: Hepatocellular carcinoma (HCC) patients undergoing hepatic angiography mapping prior to TARE (N=10)
- microwave ablation: percutaneous tumor ablation in patients receiving image-guided tumor ablation using MWA (n=10)
- cryoablation: cryoablation (N=10) for primary liver (HCC) or primary kidney tumors (RCC)

SUMMARY:
This is a pilot study to evaluate the feasibility, image quality, and procedural utility of a novel spectral CT technique using Canon Medical's 4D CT system during image-guided interventional oncology procedures

DETAILED DESCRIPTION:
The aims of this study are:

1. Demonstrate the feasibility of acquisition and image quality of intra-arterial spectral CT images obtained during mapping arteriography prior to trans arterial radioembolization (TARE) for liver cancer treatment.

   1. Assess the procedural utility of Spectral CT images as part of the TARE workflow, such as hepatopulmonary shunt fraction estimation, lesion identification, prediction of tumor: normal liver (T:N) dose ratio, and dose distribution
   2. Investigate the feasibility, safety, and image quality of Spectral CT images obtained during tumor ablation.
2. Explore the feasibility of assessing physiologic tissue changes using Spectral CT (effective anatomic number maps)

   1. During ablation with microwave, cryoablation, and irreversible electroporation in an ex vivo model
   2. For image-guided tumor ablation, such as lesion identification, probe placement, and ablation monitoring.

ELIGIBILITY:
Inclusion criteria:

1. Age > or = 18 years
2. Tumor in an area without prior surgical or ablative therapy
3. At least 1 tumor greater than 1.5 cm in greatest diameter

Exclusion criteria:

1. Not eligible for indicated procedure.
2. BMI > 35
3. Prior surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with liver or kidney cancer being treated at VAPAHCS
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
CT image | Baseline
  Effective Dose and CTDI

SECONDARY OUTCOMES:
number | Baseline
  Number of spectral CT acquisitions per patient
time | Baseline
  Fluoroscopy Time

CONTACTS AND LOCATIONS:
Overall Officials: Sirish Kishore, MD, Principal Investigator — VA Palo Alto Health Care System
Locations (1):
- VA Palo Alto Healthcare System, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2024-08-27): https://cdn.clinicaltrials.gov/large-docs/25/NCT07303725/ICF_000.pdf